CLINICAL TRIAL: NCT04106479
Title: Do Cerebral and Renal Saturations Measured With Near-infrared Spectroscopy Correlate With Echocardiographic Markers of Perfusion and Cardiac Performance in Congenital Heart Disease?
Brief Title: NIRS in Congenital Heart Defects - Correlation With Echocardiography
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Gabriel Altit, Neonatologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2018-3823
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Congenital Heart Defect; Single-ventricle; Coarctation of Aorta; Atrioventricular Canal; Hypoplastic Left Heart; Transposition of Great Vessels; Interrupted Aortic Arch; Tricuspid Atresia; Pulmonary Atresia; Aortic Atresia; Tetralogy of Fallot
MeSH Terms: conditions — Heart Defects, Congenital; Univentricular Heart; Aortic Coarctation; Endocardial Cushion Defects; Hypoplastic Left Heart Syndrome; Transposition of Great Vessels; Tricuspid Atresia; Pulmonary Atresia; Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: NIRS evaluation — NIRS will be used for measurement of cerebral and renal saturation.

SUMMARY:
Neonatal patients with congenital heart defects (CHD) have changing physiology in the context of transitional period. Patients with CHD are at risk of low perfusion status or abnormal pulmonary blood flow. Near infrared spectroscopy has been used in neonatal intensive care units (NICU) to measure end-organ perfusion. The investigator plan on monitoring newborns with CHD admitted to the NICU with NIRS and echocardiography during the first week of life and correlate measures of perfusion from Dopplers to cerebral and renal NIRS.

DETAILED DESCRIPTION:
Near infrared spectroscopy (NIRS) is a noninvasive technology that uses infrared light to measure Oxygen levels in tissue or organs. However, the use of this monitoring tool has not been the standard of care in the immediate post-natal life. The investigator wish to study this way of monitoring Oxygen, which consists of using a sticker on the skin of the forehead and the skin of the abdomen to continuously monitor the Oxygen content of the brain and the kidneys and compare NIRS values in the CHD population to echocardiographic measures of blood flow and heart function to see if/how this simple, non-invasive tool could help us to closely monitor Oxygen in babies with CHD.

The NIRS probe (sticker) will be put on the side of the abdomen (the flank to monitor the kidney saturation of oxygen) and on the forehead (to monitor the brain saturation of oxygen) for 7 days or until the baby is discharged home, has a procedure in cath-lab or has surgery. An echocardiography will take place daily (for up to 7 days, or up to discharge, or up to cardiac intervention) during the day and should last about 15- 20 minutes. Newborns will be recruited during the fetal consultation with the cardiologist or neonatologist; or will be recruited during their neonatal admission. Only newborns admitted to the NICU will be eligible to the study.

The investigator would like to better understand the way babies with cardiac conditions transition once they are born and into their first week of life. During that important time, there are a lot of changes that can impact the cardiac adaptation: vessels in the lungs that relax, vessels in the body that contract. Echocardiography and NIRS may help us better appreciate these changes by evaluating the delivery of oxygen to organs. Echocardiography may reveal some information about this adaptation by looking at the cardiac performance by ultrasound and blood flow patterns.

Approximately 100 participants from this hospital will take part in this study.

ELIGIBILITY:
Inclusion Criteria:

A prospective study will be conducted of all newborns with tetralogy of fallot, trucus arteriosus, D-transposition of great arteries, PS, AS, coarctation of the aorta, DILV, AVC, DORV, HLHS, TA and PAIVS consecutively admitted at our institution (Montreal Children's Hospital) neonatal intensive care unit (NICU) from January 2018 to January 2020. Patients with CHD will be compared to a control population of term infants admitted and monitored in the NICU with antenatal suspicion of coarctation, ruled-out postnatally.

Exclusion Criteria:

Patients will be excluded if premature less than 34 weeks of estimated gestational age (GA) at birth or if parents do not consent. Parental consent can be withdrawn at any time during the study.

Ages: 0 Days to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All newborns with tetralogy of fallot, truncus arteriosus, D-transposition of great arteries, PS, AS, coarctation of the aorta, DILV, AVC, DORV, HLHS, TA and PAIVS consecutively admitted at our institution (Montreal Children's Hospital) neonatal intensive care unit (NICU) from January 2018 to January 2020.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-11 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between cerebral saturation and ACA doppler | Measures from Day 0 to Day7
Correlation between aortic doppler and renal NIRS measures | Measures from Day 0 to Day7

SECONDARY OUTCOMES:
Correlation between LV performance by STE and Csat and Rsat by NIRs | Measures from Day 0 to Day7

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Altit, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Mcgill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Altit G, Bhombal S, Chock VY. End-organ saturations correlate with aortic blood flow estimates by echocardiography in the extremely premature newborn - an observational cohort study. BMC Pediatr. 2021 Jul 12;21(1):312. doi: 10.1186/s12887-021-02790-1. PMID 34253175